CLINICAL TRIAL: NCT04857736
Title: A Diagnostic Test Study of Characteristic Sound Waves in Radial Artery During Menstruation in Healthy Female College Students
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, dean of orthopedic department, Qianfoshan Hospital
Other Study IDs: SFUYIN-02
Record Dates: First submitted 2021-03-10; First posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Menstruation; Radial Artery
Keywords: Menstruation; Healthy Female College Students; Diagnostic Test; Radial Artery; sound waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trial group: 62 healthy female college students during menstruation: The pulse sound waves of three parts and five layers of each of the two hands of 62 healthy female college students during menstruation will be collected by the"Pulse Detection System of Sound Waves".
- Control group :62 healthy female college students during non-menstrual period: The pulse sound waves of three parts and five layers of each of the two hands of 62 healthy female college students during non-menstrual period will be collected by the "Pulse Detection System of Sound Waves".

SUMMARY:
Pulse diagnosis is an important method to judge the status of patients in the process of diagnosis and treatment of traditional Chinese medicine. At present, the commonly used site of pulse diagnosis is the radial artery, which is divided into "cun""guan" and "chi".During menstruation, the secretion of estrogen and progesterone drops to the lowest level. On the 7th day of menstruation in the proliferative period, the secretion of estrogen increases rapidly and rises to the first peak before ovulation. In the mid-secretory period, the secretion of estrogen rises to another peak, and the secretion of progesterone also reaches the highest peak. The state of the endometrium during non-menstrual period can be significantly different from the state of exfoliation and necrosis during menstruation. There are obvious differences in hormone levels and endometrial state and thickness in menstrual period and secretory period, especially in the middle and late secretion period, which affects the blood laminar flow of the uterine wall and is reflected in the acoustic information of the radial artery. Therefore, exploring the pulse manifestation of physiological menstruation can be expected to lay the foundation for assisting the diagnosis of pathological menstruation and endometrial diseases.

Our team found that there are low-frequency sound waves in the radial artery, which carry the physiological and pathological information of the organs in the body, and developed a "Pulse Detection System of Sound Waves ". Previous projects have explored the abnormal sound waves of radial artery in patients with sequelae of cerebral infarction, stable coronary heart disease, chronic gastritis, neck-shoulder syndrome, liver cirrhosis and other diseases and achieved certain results.

Therefore, in this study, the "Pulse Detection System of Sound Waves " will be used to collect the sound waves in the radial artery of 62 healthy female college students during menstruation and non-menstrual period within the same menstrual cycle , and researchers will carry on the frequency spectrum analysis and wavelet analysis to extract the pulse features. A diagnostic test was carried out by researchers to calculate the sensitivity and specificity of the "Sonic Pulse Detection System" in menstrual diagnosis. This study will verify the efficacy of pulse diagnosis of traditional Chinese medicine in the diagnosis of menstruation and lay a foundation for the diagnosis of pathological menstruation and endometrial diseases .

ELIGIBILITY:
Inclusion Criteria:

Trial group:

1. Research period: March 9, 2021 to March 9, 2022;
2. Research site: The First Affiliated Hospital of Shandong First Medical University;
3. Healthy female college students with normal menstruation of Shandong University of Traditional Chinese Medicine;
4. Menstrual period in the same menstrual cycle: Days 2nd-4th of the menstrual cycle;
5. Unmarried female college students aged 18-27 years old;
6. Female college students with informed consent to accept this pulse collection.

Control group:

1. Research period: March 9, 2021 to March 9, 2022;
2. Research site: The First Affiliated Hospital of Shandong First Medical University;
3. Healthy female college students with normal menstruation of Shandong University of Traditional Chinese Medicine;
4. Non-menstrual periods of the same menstrual cycle: Days 20th-28th of the menstrual cycle;
5. Unmarried female college students aged 18-27 years old;
6. Female college students with informed consent to accept this pulse collection.

Exclusion Criteria:

1. Special menstruation: bimonthly menstruation, seasonal menstruation, annual menstruation and latent menstruation;
2. Pregnant or lactating women;
3. Ovulation period: generally on the 14th day before menstruation and three days before it and four days after it;
4. Those with dysmenorrhea;
5. Those with severe diseases;
6. Patients with uterine or adjacent organ tissue diseases, including gynecological diseases, and diseases of waist, pelvis, colon and urinary system；
7. Those with infectious diseases;
8. Those who are not easy to collect pulse manifestation such as pulse on back of wrist and oblique-running pulse;
9. Incomplete information that affects the judgment of results due to subjective or objective reasons;
10. Those with tremor of limbs.

Ages: 18 Years to 27 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Healthy female college students with normal menstruation of Shandong University of Traditional Chinese Medicine.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-03-09 (Estimated); Study Completion 2022-03-09 (Estimated)

PRIMARY OUTCOMES:
Frequencies of abnormal sound waves in the pulses. | The data will be collected, analyzed and calculated in about 7 days.
  Using Pulse Detection System of Sound Waves (PDSSW) to collect the pulse waves of both hands. The percentage% of Frequencies of abnormal sound waves in the pulse will be calculated.
The Changes of sound waves in the pulses. | The discovery of characteristic sound waves may take 3 months.
  The Changes of sound waves at different Hertz(Hz) frequencies and SMPL(Units of cool edit amplitude) amplitudes will be compared between menstrual period and non-menstrual period of healthy female college students.
Diagnostic test | Diagnostic tests may take about 1 month.
  The percentage(%) of specificity, sensitivity, positive likelihood ratio and negative likelihood ratio of the "Pulse Detection System of Sound Waves" in the diagnosis of the menstrual period of healthy female college students.
Sound waves analysis | 1 month.
  The Hertz (Hz) of the different segments of the sound waves in Wavelet transform.
  The Hertz (Hz) of the different layers of the sound waves in Hilbert-Huang. The SMPL amplitudes of the sound waves in Discrete Fourier Transform. The sampEn of sound waves in Sample Entropy.

CONTACTS AND LOCATIONS:
Overall Officials: Lucheng Song, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Background] Lee JHS, Cheng EOL, Choi KM, Ngu SF, Cheung RYK; Hong Kong College of Obstetricians and Gynaecologists. 2020 Hong Kong College of Obstetricians and Gynaecologists guideline on investigations of premenopausal women with abnormal uterine bleeding. Hong Kong Med J. 2020 Dec;26(6):520-525. doi: 10.12809/hkmj208897. PMID 33350964
- [Background] Ullrich ND, Koschak A, MacLeod KT. Oestrogen directly inhibits the cardiovascular L-type Ca2+ channel Cav1.2. Biochem Biophys Res Commun. 2007 Sep 21;361(2):522-7. doi: 10.1016/j.bbrc.2007.07.054. Epub 2007 Jul 23. PMID 17662243
- [Background] Lawlor DA, Timpson N, Ebrahim S, Day IN, Smith GD. The association of oestrogen receptor alpha-haplotypes with cardiovascular risk factors in the British Women's Heart and Health Study. Eur Heart J. 2006 Jul;27(13):1597-604. doi: 10.1093/eurheartj/ehi833. Epub 2006 Mar 21. PMID 16551651
- [Background] Kim J, Bae JH, Ku B, Yim MH, Ang L, Kim H, Jeon YJ. A comparative study of the radial pulse between primary dysmenorrhea patients and healthy subjects during the menstrual phase. Sci Rep. 2019 Jul 4;9(1):9716. doi: 10.1038/s41598-019-46066-2. PMID 31273265
- [Background] Kim JU, Jeon YJ, Kim YM, Lee HJ, Kim JY. Novel diagnostic model for the deficient and excess pulse qualities. Evid Based Complement Alternat Med. 2012;2012:563958. doi: 10.1155/2012/563958. Epub 2011 Sep 5. PMID 21941587
- [Background] Minson CT, Halliwill JR, Young TM, Joyner MJ. Influence of the menstrual cycle on sympathetic activity, baroreflex sensitivity, and vascular transduction in young women. Circulation. 2000 Feb 29;101(8):862-8. doi: 10.1161/01.cir.101.8.862. PMID 10694525
- [Background] Su SY, Wei CC, Hsieh CL, Tsao JY, Li TC, Lin TH, Chang HH, Lo LC. Influence of menstrual cycle on pulse pressure waveforms measured from the radial artery in biphasic healthy women. J Altern Complement Med. 2009 Jun;15(6):645-52. doi: 10.1089/acm.2008.0022. PMID 19480601
- [Background] Tada Y, Yoshizaki T, Tomata Y, Yokoyama Y, Sunami A, Hida A, Kawano Y. The Impact of Menstrual Cycle Phases on Cardiac Autonomic Nervous System Activity: An Observational Study Considering Lifestyle (Diet, Physical Activity, and Sleep) among Female College Students. J Nutr Sci Vitaminol (Tokyo). 2017;63(4):249-255. doi: 10.3177/jnsv.63.249. PMID 28978872
- [Background] Maybin JA, Critchley HO. Menstrual physiology: implications for endometrial pathology and beyond. Hum Reprod Update. 2015 Nov-Dec;21(6):748-61. doi: 10.1093/humupd/dmv038. Epub 2015 Aug 7. PMID 26253932